CLINICAL TRIAL: NCT04074954
Title: A (Prospective/Pilot) Study Evaluating the Effect of Cataract Surgery on the Daily Activity Levels of Elderly Patients
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled
Sponsor: University of Pikeville (Other)
Responsible Party: Sponsor
Other Study IDs: CataractStudy1
Record Dates: First submitted 2019-08-22; First posted 2019-08-30 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2022-08

CONDITIONS: Cataract; Diabetes; Hypertension; Obesity; Vision Disability
MeSH Terms: conditions — Cataract; Diabetes Mellitus; Hypertension; Obesity; Vision Disorders | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cataracts present, no surgery: Adult patients undergoing bilateral cataract surgery
- Cataracts present, yes surgery: adult patients who have cataracts but are not undergoing cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Patients will receive cataract surgery
  Groups: Cataracts present, yes surgery

SUMMARY:
To evaluate the effect of bilateral cataract surgery with intraocular lens implantation on the daily activity levels of elderly patients.

DETAILED DESCRIPTION:
Cataract formation is a natural aging process that can be influenced by environmental factors such as exposure to ultra violet light and diet. Additionally, metabolic disorders, such as diabetes can lead to an earlier development of cataracts. As cataracts develop, a patient's vision can be affected. Reduced vision can limit activities of daily living and may even reduce a patient's mobility. When this occurs, cataract surgery should be considered to help restore a patient's vision. With the obesity and diabetic epidemic, proper diet and exercise is a major health initiative to control these diseases. If a patient's mobility is reduced as a result of poor vision - their ability to achieve adequate daily physical activity may also be effected. It is thought that improvement in vision may increase their activity levels and help combat these health issues. This study will investigate the activity level of patients before and after undergoing cataract surgery to determine how improved vision quality from removal of the natural lens inside the eye and replacement with an artificial intraocular lens effects their activity level.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral cataract extraction by phacoemulisficatin with intraocular lens implantation and a planned bilateral distance vision target or patients with bilateral cataracts who are not having cataract surgery
* Patients aged 60 years old or older
* Best corrected visual acuity worse than 20/20 in each eye (meaning 20/25 or worse)
* Non-comanged patients

Exclusion Criteria:

* Greater than 0.76 D pre-operative corneal cylinder, if having cataract surgery without a planned astigmatism correction (I.e Limbal relaxing incision or Toric intraocular lens)
* Planned implantation of a multifocal intraocular lens
* Visual field defect which may reduce mobility
* Wheel chair bound patients
* Reduced vision from an ocular disease other than cataracts
* Patients with significant dementia who are not able to fully comprehend the informed consent

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing bilateral cataract surgery and adult patients who have cataracts but are not undergoing cataract. Consecutive patients based on the inclusion criteria will be selected for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-23 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Amount of activity conducted by the patient before receiving surgery | 10 days prior to surgery
  Measured by a wrist activity tracker
Amount of activity conducted by the patient after receiving surgery | 10 days after surgery
  Measured by a wrist activity tracker

CONTACTS AND LOCATIONS:
Overall Officials: Kelley E Sedlock, OD, Principal Investigator — University of Pikeville
Locations (1):
- Bennett and Bloom Eye Centers, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT04074954/Prot_000.pdf